CLINICAL TRIAL: NCT05227443
Title: Effects of Different Exercise Training Programs on the Functional Performance in Fibrosing Interstitial Lung Diseases
Brief Title: Effects of Exercise Training on Respiratory Performance in Patients With Fibrosing Interstitial Lung Diseases
Acronym: ET-fILD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Hanaa Shafiek, Assistant professor, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0201313
Record Dates: First submitted 2021-12-22; First posted 2022-02-07 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Lung Diseases; Interstitial Lung Disease; Fibrosis Lung
MeSH Terms: conditions — Lung Diseases; Lung Diseases, Interstitial; Pulmonary Fibrosis | interventions — Respiration; Exercise

STUDY DESIGN:
Intervention Model Description: The current study has 2 groups of patients subjected to 2 different modalities of aerobic exercise training and a control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): The control group did not receive exercise training and the participants were informed to complete their medications provided by the treating physician.
- Lower limb (LL) exercise training (Active Comparator): All the participants in this modality of training were subjected to only lower limbs aerobic exercise training.
  Interventions: Procedure: Exercise aerobic training
- Upper, lower and breathing (ULB) exercise training (Active Comparator): All the participants in this modality of training were subjected to upper and lower limb aerobic exercise training as well as breathing training.
  Interventions: Procedure: Upper, lower and breathing (ULB) exercise

INTERVENTIONS:
Procedure: Exercise aerobic training — It is a procedure that is in the form of exercise training as a part of rehabilitation. The patients were subjected to 3 supervised sessions of exercise training / week for a total duration of 6 weeks. The form of training was aerobic intensity exercise that lasts for 15 minutes of continuous exercise. In this intervention, the investigators provide only lower limbs training exercises.
  Other Names: Lower limbs (LL) training
  Arms: Lower limb (LL) exercise training
Procedure: Upper, lower and breathing (ULB) exercise — It is a procedure that is in the form of exercise training as a part of rehabilitation. The patients were subjected to 3 supervised sessions of exercise training / week for a total duration of 6 weeks. The form of training was aerobic intensity exercise that lasts for 15 minutes of continuous exercise. In this intervention, the investigators provide lower and upper limbs training exercises as well as breathing exercises.
  Arms: Upper, lower and breathing (ULB) exercise training

SUMMARY:
The current study recruited patients with fibrosing interstitial lung diseases (f-ILD) whatever was the underlying pathology. The investigators aimed to compare the effects of aerobic exercises for lower limbs (LL) versus upper limbs, lower limbs, and breathing exercises (ULB) on the peak exercise measurements that was measured using cardiopulmonary exercise testing (CPET), dyspnea and health related quality of life assessment in this group of patients.

DETAILED DESCRIPTION:
The investigators conducted a case-control study with a follow up after 6 weeks (short term). All the participants on recruited were evaluated clinically. A high resolution computed tomography (HRCT) scan of the chest was performed to confirm the diagnosis of f-ILD as well as a spirometry. All the patients were subjected to cardiopulmonary exercise testing (CPET), 6-minute walk test (6-MWT), evaluation of dyspnea using mMRC dyspnea scale, and evaluation of health related quality of life using St. George's Respiratory Questionnaire (SGRQ). The control group were followed up by telephone calls. The intervention groups (LL and ULB) were subjected randomly to aerobic exercise training for 6 weeks. After termination of all the session, the patients were re-evaluated clinically and objectively using CPET, 6-MWT, mMRC and SGRQ. Also, we evaluated the outcome of the patients (control and intervention groups) as those who died or reported exacerbation of the underlying disease were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged ≥ 18 years.
* Fibrosis interstitial lung diseases (f-ILDs) diagnosed based on HRCT radiological features.
* Restrictive or mixed pattern in forced spirometry test

Exclusion Criteria:

* Motor disabilities
* Cardiovascular diseases (as acute heart failure, unstable angina or recent myocardial infarction)
* Cognitive impairments
* History of cerebrovascular accident
* Active cancer
* Life expectancy less than 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Maximum oxygen consumption | 6 weeks
  Cardiopulmonary exercise testing (CPET) was used to assess the improvement of maximum oxygen consumption.
Quality of life evaluation | 6 weeks
  St. George's Respiratory Questionnaire (SGRQ) was used to assess the health related quality of life. SGRS constitutes 50 items and the score ranging from 0 to 100, with higher scores indicating more limitations.

SECONDARY OUTCOMES:
Dyspnea | 6 weeks
  mMRC dyspnea scale (ranging from 0 (the best) - 4 ( the worst) was used to evaluate the improvement of dyspnea.
Resting oxygen saturation | 6 weeks
  Pulse oximeter was used to assess the change in oxygen saturation (SaO2) at rest after termination of exercise sessions. SaO2 is presented as percentage (%).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
We are planning to share IPD but until now we did not decided as we need to talk with all the researchers conducted the trial before it is available for the public. For the time being, the data is available on request from the principal investigator.